CLINICAL TRIAL: NCT03243279
Title: Role of Preoperative Baroreflex Sensitivity on Major Outcomes After Cardiothoracic Surgery
Brief Title: BRS and Outcomes in Cardiothoracic Surgery
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00083136
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative; Atrial Fibrillation; Cognitive Dysfunction
MeSH Terms: conditions — Pain, Postoperative; Atrial Fibrillation; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical: No interventions. Patients undergoing cardiothoracic surgery will be assessed for baroreflex sensitivity and the outcomes of interest.

SUMMARY:
The purpose of this study is to determine whether baroreceptor sensitivity (the ability of your body to change your heart rate and/or blood pressure in response to a situation) has any effect on how likely you are to suffer certain events after heart or lung surgery. The postoperative events that the investigators will be studying are pain after surgery, atrial fibrillation (an irregular heart rhythm), and cognitive dysfunction (a decline in mental abilities).

DETAILED DESCRIPTION:
The purpose of this study is to determine if preoperative baroreceptor sensitivity (BRS) correlates with major outcomes after cardiac and thoracic surgery, including acute and chronic pain, atrial arrhythmias, and cognitive function. To test this hypothesis, approximately 95 patients will be enrolled, and spontaneous baroreceptor sensitivity will be measured prior to surgery as well as immediately postoperatively. Outcomes will include acute pain using the numeric rating scale, Brief Pain Inventory, and Gracely Box Scale administered preoperatively, on postoperative days 1 and 2 and by phone at 6-weeks postoperatively. Chronic pain will be assessed at 6-month follow-up visit via hyperalgesia testing using Von Frey filaments. Postoperative atrial arrhythmias will be assessed by review of postoperative telemetry, the electronic medical record, and ECG performed prior to discharge. Finally, cognitive function will be assess via Mini-Mental State examination administered preoperative and at the 6-month follow-up visit. Association between BRS and the outcomes of interest will be tested with regression models adjusted for appropriate covariates. Significance threshold alpha will be adjusted for the number of statistical tests using the Bonferroni correction. Our hypothesis is that patients with impaired preoperative BRS will have an increased incidence of acute and chronic postoperative pain, atrial fibrillation, and cognitive decline after surgery.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Undergoing cardiac (coronary artery bypass grafting [CABG], CABG + valve, or valve only) or thoracic (video-assisted thoracoscopic [VATS] approach to lobectomy) surgery

Exclusion Criteria:

* Any preexisting pain condition (defined as pain of >=3 months duration prior to enrollment)
* Pain at the time of enrollment interview
* Need for preoperative analgesics
* Preexisting chronic or paroxysmal atrial fibrillation
* Preexisting atrial or ventricular arrhythmia
* Need for preoperative anti-arrhythmic medication
* History of symptomatic cerebrovascular disease (e.g., prior stroke) with residual deficits
* Alcoholism (>2 drinks/day)
* Psychiatric illness (any clinical diagnosis requiring therapy)
* Drug abuse (any illicit drug use in the preceding 3 months before surgery)
* Hepatic insufficiency (liver function tests > 1.5 times the upper limit of normal)
* Severe pulmonary insufficiency (home oxygen)
* Renal failure (serum creatinine >2.0 mg/dL)
* Non-English speaking
* Unable to read
* Participants who score <24 on baseline Mini Mental State examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting for cardiac and thoracic surgery at Duke University Hospital, a quaternary referral center
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Baseline baroreflex sensitivity | 30 min
  Non-invasive BRS testing with BIOPAC MP160

SECONDARY OUTCOMES:
Postoperative day (POD) 1 baroreflex sensitivity | 30 min
  Non-invasive BRS testing with BIOPAC MP160
POD 2 baroreflex sensitivity | 30 min
  Non-invasive BRS testing with BIOPAC MP160
6 month baroreflex sensitivity | 6 months
  Non-invasive BRS testing with BIOPAC MP160
Acute postoperative pain as assessed by the numeric rating scale (NRS) - 24h | 24 hours
  Median NRS pain score in the first 24h after surgery
Acute postoperative pain as assessed by the numeric rating scale (NRS) - 48h | 48 hours
  Median NRS pain score in the second 24h after surgery
Acute postoperative pain as assessed by the Gracely Box Scale (GBS) - POD1 | 15 min
  GBS survey on POD 1
Acute postoperative pain as assessed by the Gracely Box Scale (GBS) - POD2 | 15 min
  GBS survey on POD 2
Acute postoperative pain as assessed by the Gracely Box Scale (GBS) - 6 mo | 6 months
  GBS survey at 6 month follow-up visit
Chronic pain as assessed by the change in Brief Pain Inventory score | Baseline, 6 months
  Change from baseline to 6 months postoperatively
Hyperalgesia | 6 months
  Nociceptive threshold as assessed by Von Frey filament testing at 6 month follow-up
Area of hyperalgesia or allodynia | 6 months
  Area surrounding operative incision as assessed by Von Frey filament testing at 6 month follow-up
Postoperative atrial fibrillation | 6 weeks
  Chart review assessment of the occurrence of postoperative atrial fibrillation during hospitalization and up to 6 weeks postoperatively
Postoperative cognitive change | Baseline, 6 months
  Change from baseline to 6 months in the Mini Mental Status Exam score
Baseline psychological distress | 15 min
  As assessed by the Brief Symptom Inventory-18
6 month psychological distress | 6 months
  As assessed by the Brief Symptom Inventory-18
Baseline frailty | 10 min
  As assessed by the Modified Frailty Index

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided